CLINICAL TRIAL: NCT00163813
Title: The Early Nasojejunal Tube to Meet Energy Requirements in Intensive Care Study
Brief Title: The Early Nasojejunal Tube to Meet Energy Requirements in Intensive Care (ENTERIC) Study
Acronym: ENTERIC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bayside Health (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 232/04
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2007-02-26 (Estimated); Status verified 2005-08

CONDITIONS: Critical Illness; Malabsorption Syndromes
Keywords: Mechanically-ventilated; medical-surgical critically ill patients; reduced gastric motility
MeSH Terms: conditions — Critical Illness; Malabsorption Syndromes

INTERVENTIONS:
Procedure: Early jejunal feeding (using frictional NJ tube)
Procedure: Standard feeding (using nasogastric [NG] tube)

SUMMARY:
This is a multi-centre randomised controlled trial comparing early jejunal feeding (using a frictional nasojejunal [NJ] tube) and standard feeding in critical illness.

ELIGIBILITY:
Inclusion Criteria:

ICU patients are eligible for enrolment if they meet all of the following:

* Age > 18 years old
* In ICU for < 48 hours prior to enrolment
* Receiving invasive mechanical ventilation (through an endotracheal tube or tracheostomy, but NOT a facemask) with an anticipated need for > 48 hours of mechanical ventilation
* Receiving a continuous infusion of any one of:

  * morphine > 2 mg/hour,
  * fentanyl > 20 mcg/hour, or
  * pethidine > 20 mg/hour
* Either a single GRV > 150 mls (whilst receiving EN via a NG tube) or nasogastric drainage > 500 mls over 12 hours (whether receiving EN or not)

Exclusion Criteria:

Patients will be ineligible for enrolment if they meet any of the following:

* Previous or recent surgery which has altered the anatomy of the upper gastrointestinal tract (eg. oesophagectomy, gastrectomy, any gastric anastomosis surgery, gastroplasty, pyloroplasty, pancreaticoduodenectomy [Whipple's procedure])
* Known gastric malignancy
* Known oesophageal varices
* Current admission for peptic ulceration
* Current mechanical bowel obstruction
* Current gastrostomy, jejunostomy, or surgically-placed enteral tube in situ
* Contraindication to the use of the nose and mouth for enteral tube insertion (eg. recent facial trauma or surgery)
* Receiving nutritional support prior to ICU admission
* Severe coagulopathy (defined by platelet count < 20 and/or international normalized ratio [INR] > 4.0)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180

PRIMARY OUTCOMES:
The amount of EN delivered during the Intensive Care Unit (ICU) stay

SECONDARY OUTCOMES:
Amount of EN delivered during the first 10 days of the study
Daily cumulative proportion of EN delivered
Ventilator-associated pneumonia rate
Duration of mechanical ventilation
Duration of hospitalisation
Mortality at hospital discharge
Success rate of placement into both the small bowel, generally, and the jejunum, specifically
Complication rates (as compared to the nasogastric tube)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Davies, Principal Investigator — The Alfred
Locations (1):
- Alfred Hospital, Melbourne, Victoria, Australia